CLINICAL TRIAL: NCT06243328
Title: A Randomised Clinical Trial of the Negative Pressure Wound Therapy Versus Conventional Dressing for Pressure Ulcers Management
Brief Title: Effect of Negative Wound Pressure on P.S
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, issraa Aly, resident doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAC on PS
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Pressure Sores
MeSH Terms: conditions — Pressure Ulcer | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Masking Description: Based on determining the main outcome variable, the estimated minimum required sample size is 39 patients (13 patient in each group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional dressing (Experimental): The surface of the PU will be cleaned with normal saline and packed with sterilised gauze to cover the wound. Dressing changes will be performed once or twice daily depending on the soakage of the dressing
  Interventions: Device: negative wound pressure therapy
- negative pressure wound therapy (Experimental): We will place a nonadherent contact layer, such as Xeroform between prepared wound bed and foam then applying a contact dressing with sealling using an adhesive drape. The dressing will be connected to the machine through tubing that was connected to the canister. Continuous pressure of 200 mm Hg will be applied. The dressing will be changed three times a week.
  Interventions: Device: negative wound pressure therapy

INTERVENTIONS:
Device: negative wound pressure therapy — nonadherent contact layer, such as Xeroform between prepared wound bed and foam then applying a contact dressing with sealling using an adhesive drape. The dressing will be connected to the machine through tubing that was connected to the canister

SUMMARY:
This study will compare the NPWT using the NPD to the conventional wound dressing and specifically evaluating (i) reduction of wound surface area and depth, (ii) removal of slough and formation of granulation tissue

DETAILED DESCRIPTION:
Initial debridement of slough and necrotic tissue was performed in all patients at the time of admission and before their being allocated in a group.

it's 3 groups:

Group (A): conventional dressing :

acting by:preventing pus, the findings from the review indicate that decreasing frictional forces transmitted to the patient's skin is achieved by use of a dressing with an outer surface made from a low friction material.

The surface of the PU will be cleaned with normal saline and packed with sterilised gauze to cover the wound. Dressing changes will be performed once or twice daily depending on the soakage of the dressing.

.

Group (B), negative pressure wound therapy using the electronic-vac :

It is believed that the negative pressure assists in removal of interstitial fluid, decreasing oedema, increasing blood flow and reducing tissue bacterial levels, in addition, mechanical deformation of cells is thought to result in protein and matrix molecule synthesis, which increases the rate of cell proliferation and granulation tissue formation, this , in turn , may promote healing .

We will place a nonadherent contact layer, such as Xeroform between prepared wound bed and foam then applying a contact dressing with sealling using an adhesive drape. The dressing will be connected to the machine through tubing that was connected to the canister. Continuous pressure of 200 mm Hg will be applied. The dressing will be changed three times a week Group (C), negative pressure wound therapy using the Romo-vac: The NPD will be applied as a bedside procedure with a low-power continuous suction apparatus. We will Place nonadherent contact layer, such as Xeroform between prepared wound bed and contact dressing with sealling using an adhesive drape. The dressing will be connected to the Romo-vac which applying pressure of-60 to -125 mm Hg. The Romo-vac will be recharged every 5-6 hours and the dressing will be changed three times a week or earlier if there is a soakage/leakage

ELIGIBILITY:
Inclusion Criteria:

Stages three and four PU as defined by the National Pressure Ulcer Advisory Panel (NPUAP).

Exclusion Criteria:

* wound with necrotic tissue unlikely to tolerate debridement. Exposed Vessels, Nerves and or organs. Active bleeding. Ischemic limb. Opening into body cavity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ulcer size | 3 weeks
  measured for its greatest length ,depth and width with flexigrid Opsite.

CONTACTS AND LOCATIONS:
Overall Officials: assem hussien, professor, Principal Investigator — Assiut University

REFERENCES:
- [Background] Avsar P, Moore Z, Patton D. Dressings for preventing pressure ulcers: how do they work? J Wound Care. 2021 Jan 2;30(1):33-39. doi: 10.12968/jowc.2021.30.1.33. PMID 33439083
- [Background] Srivastava RN, Dwivedi MK, Bhagat AK, Raj S, Agarwal R, Chandra A. A non-randomised, controlled clinical trial of an innovative device for negative pressure wound therapy of pressure ulcers in traumatic paraplegia patients. Int Wound J. 2016 Jun;13(3):343-8. doi: 10.1111/iwj.12309. Epub 2014 Jun 3. PMID 24894079
- [Background] Lesiak AC, Shafritz AB. Negative-pressure wound therapy. J Hand Surg Am. 2013 Sep;38(9):1828-32. doi: 10.1016/j.jhsa.2013.04.029. Epub 2013 Jun 25. No abstract available. PMID 23809469